CLINICAL TRIAL: NCT02375750
Title: Surgical Treatment of Peri-implantitis Lesions, With or Without the Placement of a Bone Substitute and a Collagen Membrane. A Randomized Clinical Trial
Brief Title: Treatment of Peri-implantitis Lesions by Using Biomaterial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS13530231
Record Dates: First submitted 2014-07-07; First posted 2015-03-03 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GBO and GBG (Experimental): 0.2 g-0,5 g GBO and 1 GBG once after decontamination of implant surface
  Interventions: Device: GBO and GBG
- Standard treatment (Active Comparator): Decontamination of surface of implant
  Interventions: Other: Standard treatment

INTERVENTIONS:
Device: GBO and GBG — Application of GBO and GBG to the defect fill after removal of chronic inflammatory tissue and decontamination of the surface of implant
  Arms: GBO and GBG
Other: Standard treatment — Removal of chronic inflammatory tissue using titanium curettes and a rotary titanium brush; Implant Surface decontamination and closure by suturing
  Arms: Standard treatment

SUMMARY:
The primary objective of the study is to proof the successful use of Geistlich Bio-Oss® and Geistlich Bio-Gide® (already registered medical devices) in bony peri-implant defects due to peri-implantitis disease.

DETAILED DESCRIPTION:
Patient who will considered eligible at the screening visit will undergo surgical treatment procedure within 2 weeks. At the day of the surgery the patients will be randomized into the 2 treatment groups.

The subjects will be then prescribed postoperative antibiotics (Azitromax 500 mg day one and 250 mg day 2-4).

Post-operative pain will be controlled with Ibuprofen (400mg x 3) for two days to all subjects. Subjects will rinse twice daily with Chlorhexidine mouth rinse and use modified oral hygiene procedures during the first 5 weeks of healing. Subjects will receive professional prophylaxis as required.

Subjects will be instructed on appropriate oral hygiene throughout the study and will be given appropriate oral hygiene instructions. Instructions on post-operative care will be repeated at each visit. In particular the following points have to be covered during the first month after surgery: Chlorhexidine rinses, avoidance of brushing, usage of interdental cleaning devices, avoidance of chewing on or trauma to the treated area. In addition subjects will be instructed not to smoke more than 10 cigarettes per day during the entire study period and not to consume alcohol during antibiotic therapy.

Sutures will be removed after 14 days. Photos will be taken during the whole study to document the healing process.

Further follow up visits will be scheduled 6 weeks and 3,6,9,12 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* Presence of peri-implantitis
* A peri-implant intraosseous defect with at least 3 mm defect depth as seen on an intraoral radiograph.
* Clinically a probing depth ≥ 5 mm combined with bleeding and/or pus should be present at the site.
* During surgical exploration an intraosseous component of at least 3 mm at the deepest point must be present.
* The defect should have a minimum of 3 osseous walls (a circumference of the osseous defect of at least 270 degrees). Only 3 and 4 wall intraosseous defects will be included.
* Implants included in the study must have been in function for more than 12 months.
* Ability to fully understand the nature of the proposed surgery and ability to sign an Ethics Committee-approved informed consent form

Exclusion Criteria:

* Subjects with diabetes mellitus (HbA1c > 7.0)
* Subjects taking prednisone or other anti-inflammatory prescription drug
* Subjects taking medications known to have effects on gingival growth
* If the same patient has more than one defect meeting the inclusion criteria, only one such defect will be included in the study
* General contraindications for dental and/or surgical treatments
* Smokers (> 10 cigarettes per day).
* Pregnant or lactating women
* Allergy to collagen
* Inability to consent for participation in the study and/or to accept the proposed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-09; Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in the dimensions of the bone defect | 6 months, 1 year

SECONDARY OUTCOMES:
Change in pocket depth | 3 months,6months, 9 months,12months
Change in gingival inflammation | 3 months,6months, 9 months,12months
Changes in recession of the mucosal margin | 3 months,6months, 9 months,12months
Subject satisfaction with the outcome at the study end | 12months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Renvert, Professor, Principal Investigator — Department of Health Sciences, Kristianstad University
Locations (1):
- Kristianstad University, Department of Health Sciences, Kristianstad, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Renvert S, Giovannoli JL, Rinke S. The efficacy of reconstructive therapy in the surgical management of peri-implantitis: A 3-year follow-up of a randomized clinical trial. J Clin Periodontol. 2024 Oct;51(10):1267-1276. doi: 10.1111/jcpe.14049. Epub 2024 Jul 17. PMID 39020503
- [Derived] Renvert S, Giovannoli JL, Roos-Jansaker AM, Rinke S. Surgical treatment of peri-implantitis with or without a deproteinized bovine bone mineral and a native bilayer collagen membrane: A randomized clinical trial. J Clin Periodontol. 2021 Oct;48(10):1312-1321. doi: 10.1111/jcpe.13513. Epub 2021 Jul 29. PMID 34169551